CLINICAL TRIAL: NCT01952808
Title: Healthy Immigrant Families: Working Together To Move More and To Eat Well
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Irene G. Sia, M.D., Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13-003408
Record Dates: First submitted 2013-09-24; First posted 2013-09-30 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Immigrant Physical Activity and Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Participants randomly assigned to this group will receive the intervention immediately.
  Interventions: Behavioral: Face-to-face family mentoring and education sessions; Behavioral: Telephone follow-up
- Control Group (No Intervention): Participants randomly assigned to this group will not receive the intervention until one year after enrollment.

INTERVENTIONS:
Behavioral: Face-to-face family mentoring and education sessions — A total of 13 home visits will be completed over a 6 month period. In addition to an introductory/orientation visit, 12 home visits will consist of family mentoring/educational sessions focused on physical activity and healthy nutrition.
  Arms: Intervention Group
Behavioral: Telephone follow-up — During months 7-12, a total of up to 12 phone calls will be completed. Follow-up calls will consist of a progress report from families on physical activity and healthy diet progress/goals, along with brief content follow-up and re-enforcement points from the 12 intervention sessions.
  Arms: Intervention Group

SUMMARY:
This project will broadly explore the efficacy of community participation in the design and implementation of an intervention to improve physical activity and nutrition among immigrant and refugee (Hispanic, Somali, Sudanese, Cambodian) families in Rochester, Minnesota

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 11 years old
* Reside in a household with at least one adult and one child (11-18)
* Not planning to move from the area over the next two years
* Willing and able to participate in all aspects of the study
* Willingness to provide oral informed consent
* Hispanic, Sudanese, Somali
* Residing in Rochester, MN

Exclusion Criteria:

* Self-reported pregnancy
* Self-reported insulin-dependent diabetes
* Self-reported diagnosis of cancer within the past 3 years
* Answer of "yes" to the following question: "Do you know of any reason why you should not do physical activity? For example, would it be unsafe for you to do increased physical activity because of a health problem?"

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Improved dietary quality | Baseline- 24 months
  A 24-hour dietary recall will be collected in-person from study participants at baseline and follow-up using the Automated Self-administered 24-hour Recall (ASA24) system.
Increased physical activity | Baseline- 24 months
  The KAM (Kinetic Activity Monitor) accelerometer will be used for objective physical activity assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Sia, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Wieland ML, Weis JA, Hanza MM, Meiers SJ, Patten CA, Clark MM, Sloan JA, Novotny PJ, Njeru JW, Abbenyi A, Levine JA, Goodson M, Porraz Capetillo MG, Osman A, Hared A, Nigon JA, Sia IG. Healthy immigrant families: Participatory development and baseline characteristics of a community-based physical activity and nutrition intervention. Contemp Clin Trials. 2016 Mar;47:22-31. doi: 10.1016/j.cct.2015.12.004. Epub 2015 Dec 4. PMID 26655431